CLINICAL TRIAL: NCT00178178
Title: A Placebo Controlled, Prospective, Randomized Clinical Investigation of the Efficacy of Continuous Infusion Regional Anesthetic on Postoperative Pain Following Arthroscopic Anterior Cruciate Ligament Reconstruction: A Comparison of Three Catheter Placement Positions
Brief Title: Arthroscopic Anterior Cruciate Ligament Reconstruction: A Comparison of Three Catheter Placement Positions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: BREG, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pain Catheter Study
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2015-05-18 (Estimated); Last update posted 2015-09-11 (Estimated); Status verified 2015-08

CONDITIONS: Pain, Postoperative
Keywords: anterior cruciate ligament reconstruction; Pain Care 3000; Catheter Placement; Pain; Breg, Inc
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Drug: Bupivicaine 0.5% Intraaticulary Only (Experimental): Breg Pain Care 3000 Catheter;Bupivicaine 0.5%;Intraaticular Only
  Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) intraarticularly only via Breg Pain Care 3000 Catheter
  Interventions: Device: Breg Pain Care 3000 Catheter; Drug: Bupivicaine 0.5%
- Drug: Bupivicaine 0.5% Patellar Tendon Site (Experimental): Breg Pain Care 3000 Catheter;Bupivicaine 0.5%;Patellar Tendon Site Only
  Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the patellar tendon harvest site via Breg Pain Care 3000 Catheter
  Interventions: Device: Breg Pain Care 3000 Catheter; Drug: Bupivicaine 0.5%
- Drug: Bupivicaine 0.5% Intraarticular and Patellar Tendon (Experimental): Breg Pain Care 3000 Catheter;Bupivicaine 0.5%; Intraarticular and Patellar Tendon Sites
  Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the Patellar Tendon Harvest Site and Intraarticular infusion via Breg Pain Care 3000 Catheter
  Interventions: Device: Breg Pain Care 3000 Catheter; Drug: Bupivicaine 0.5%
- Drug: Placebo (Placebo Comparator): Breg Pain Care 3000 Catheter with Placebo
  Receive liquid with no pain medication (placebo) through a catheter in one part of the operative knee via Breg Pain Care 3000 Catheter
  Interventions: Device: Breg Pain Care 3000 Catheter; Drug: Placebo

INTERVENTIONS:
Device: Breg Pain Care 3000 Catheter — Device: Breg Pain Care 3000 Catheter
Drug: Bupivicaine 0.5% — Drug: Bupivicaine 0.5 %
  Arms: Drug: Bupivicaine 0.5% Intraarticular and Patellar Tendon; Drug: Bupivicaine 0.5% Intraaticulary Only; Drug: Bupivicaine 0.5% Patellar Tendon Site
Drug: Placebo — Drug: Placebo
  Arms: Drug: Placebo

SUMMARY:
This investigation will evaluate the subjective effect on postoperative pain of three catheter placements in the knee:

1. intraarticular infusion only,
2. patellar tendon harvest site only,
3. both intraarticular and patellar tendon harvest site.

DETAILED DESCRIPTION:
There will be 96 subjects recruited into this study. Based on power analysis for repeated measures analysis of variance, the sample size required for this investigation is 24 subjects per group based on a 90% confidence interval and alpha of 0.05. There will be 24 subjects in Group 1 (intraarticular bupivicaine infusion only). There will be 24 subjects in Group 2 (patellar tendon harvest site only with bupivicaine). There will be 24 subjects in Group 3 (both intraarticular and patellar tendon harvest site with bupivicaine). There will be 24 subjects in the control, Group 4 (intraarticular infusion physiologic saline only). All patients will be recruited under the discretion of the principal investigator.

The primary outcome measure for this investigation will be the Postoperative Patient Diary. This document records patient's subjective evaluations of pain, comfort, ability to sleep, activity level and quality of life. The Postoperative Patient Diary will be administered daily on the day of surgery and each morning and each evening before the patient retires for 3 postoperative days. All pain medications taken during the 3 days of the postoperative evaluation will be recorded on the Postoperative Patient Diary.

The investigational treatment for this investigation is the use of a Pain Care 3000 continuous infusion regional anesthesia device and accepted pharmacologic modalities for the control of postoperative pain with continuous infusion of a local anesthetic agent (bupivicaine 0.5%) intraarticularly only (Group 1), at the patellar tendon harvest site (Group 2) and combined continuous infusion at the patellar tendon harvest site and intraarticular infusion (Group 3).

Patients randomly assigned to the control group (Group 4) will receive intraarticular infusion physiologic saline only.

The catheter delivers 2 cc of bupivicaine 0.5% per hour total. In patients in Group 3, with 2 catheters (1 in the patellar tendon harvest site and 1 intraarticular infusion), the catheters are connected by a "Y" connector. The dosage of bupivicaine will be split among the two sites.

The device does not allow delivery of more than 2 cc per hour. The patient cannot adjust or alter the flow rate.

A standard general anesthetic protocol will be employed at the discretion of the supervising anesthesiologist.

Prior to surgery, all patients will be instructed on both the use of the continuous infusion device and on the methods for completing the study questionnaires. Catheters will be placed at the end of the surgical procedure according to the randomization schedule. Patients will then complete the study questionnaires on the day of surgery and on three consecutive days following surgery.

The clinical evaluation will last 3 postoperative days. During the postoperative period, sufficient additional pain medications will be available to all patients to sufficiently control postoperative pain.

No analgesics or local anesthetics, other than those specified should be taken during the postoperative period by any subject. Other medications such as "rescue analgesics" considered to be necessary to the patient's welfare will be given at the discretion of the principal investigator. If the medication provided is for pain relief, the patient must request it. The administration of all medication, from premedication until discharge from the hospital, must be recorded in the patient diary if it has a direct bearing on the study outcome. Any medication taken for pain following hospital discharge within the established post discharge follow up period must be recorded in the patient diary.

The investigator is responsible for assuring that there are procedures and expertise available to cope with medical emergencies that may occur during the study. In case of emergency, symptomatic treatment will be provided according to hospital routine. The reason for the emergency may constitute a serious adverse event.

After surgery, a patient would be discontinued from the study if it is discovered that they show a previously unrecognized allergy to the medication (bupivicaine). This would be rare. If it occurs, the catheter would be immediately removed, thus ending the infusion of the medication and the patient would no longer participate in the study.

Standard of Care Procedures:

Opioid based analgesics or their derivatives have been the standard of care in managing postoperative pain for this procedure. These medications have been administered orally, intramuscularly, or intravenously. There is no difference in the surgical procedure except for the insertion of the catheter at the surgical site upon closure of the surgical wound. All patients will receive Toradol 30 mg parenterally q6h x2, followed by Toradol 10 mg PO QID for 3 days. This anti-inflammatory has an analgesic effect and is not used prn. Any narcotic is used only as needed and the use of this will be tracked for this study.

All patients (including those in the study) will be kept in the hospital overnight following surgery and will receive a patient controlled analgesia (PCA) device for intravenous administration of morphine through the night of the hospital stay. Morphine usage during this period will be recorded.

Patients undergoing this knee surgery are admitted to the 23 hour unit, stay overnight, and are discharged the following morning usually before 10:00 am. This is the standard of care and will be the same for those participating in the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject symptoms

  1. Daily pain
  2. Pain restricts work, recreation and/or activities of daily living (ADL)
* Cognitive function sufficient to understand protocol and to complete subject diary or other analysis tools employed.
* Must read, write, and understand the English language.
* American Society of Anesthesiologists (ASA) risk 1 or 2
* Gender - Both
* Age 15 - 65 years (parental consent will be obtained on all subjects under age 18).
* Provided written informed consent

Exclusion Criteria:

* Neuropathic joint
* Remote source of ongoing sepsis
* Severe vascular disease
* Any medical condition precluding safe anesthesia, surgery, or rehabilitation
* Comorbid conditions preventing full functional activity or which require continuous use of pain medication.
* A known history of allergy, sensitivity, or any other form of reaction to local anesthetics of the amide type, acetaminophen, or opioids.
* Suspected inability to comply with study procedures, including language difficulties or medical history and/or concomitant disease, as judged by the investigator.
* A neurological and/or vascular condition which may affect the outcome of the procedure.
* Receiving regular treatment with analgesics, sedatives, or any other medication with central nervous system effects.
* Tendency to bleed
* Women who are pregnant or are not practicing medically acceptable contraception (a pregnancy test is used pre-operatively as part of standard of care).
* Participation in other clinical studies during this study or in the 14 days prior to admission to this study.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2005-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D Bronstein, MD, Principal Investigator — University of Rochester
Locations (1):
- Strong Memorial Hospital, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intraarticulary Only: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) intraarticularly only via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Patellar Tendon Harvest Site Only: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the patellar tendon harvest site via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Patellar Tendon Harvest Site and Intraarticular: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the Patellar Tendon Harvest Site and Intraarticular infusion via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Placebo: Receive liquid with no pain medication (placebo) through a catheter in one part of the operative knee via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
Period: Overall Study
Arm/Group | Intraarticulary Only | Patellar Tendon Harvest Site Only | Patellar Tendon Harvest Site and Intraarticular | Placebo
Started | 24 | 24 | 24 | 24
Completed | 24 | 24 | 24 | 24
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Drug: Intraarticularly Only: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) intraarticularly only via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Drug: Patellar Tendon Harvest Site Only: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the patellar tendon harvest site via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Drug: Patellar Tendon Harvest Site and Intraarticular: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) at the Patellar Tendon Harvest Site and Intraarticular infusion via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Placebo Comparator: Receive liquid with no pain medication (placebo) through a catheter in one part of the operative knee via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
- Total: Total of all reporting groups
Arm/Group | Drug: Intraarticularly Only | Drug: Patellar Tendon Harvest Site Only | Drug: Patellar Tendon Harvest Site and Intraarticular | Placebo Comparator | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 7 | 12 | 8 | 4 | 31
  Between 18 and 65 years | 17 | 12 | 16 | 20 | 65
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 6 | 4 | 27
  Male | 16 | 15 | 18 | 20 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 24 | 24 | 24 | 24 | 96
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 1 | 2 | 4
  White | 24 | 23 | 22 | 21 | 90
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 24 | 24 | 96

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain over the first three days post-operatively. This will be identified by the use of the Postoperative Patient Diary. This document records patient's subjective evaluations of pain, comfort, ability to sleep, activity administered daily on the day of surgery and each morning and each evening before the patient retires for 3 postoperative days. All pain medications taken during the 3 days of the postoperative evaluation will be recorded on the Postoperative Patient Diary.
Time Frame: 3 day
Measure: Number; unit: participants that experienced pain
Arm/Group | Intraarticulary Only | Patellar Tendon Harvest Site Only | Patellar Tendon Harvest Site and Intraarticular | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24
participants that experienced pain | 24 | 24 | 24 | 24

ADVERSE EVENTS:
Time Frame: 3 days
Groups:
- Intraartciularly Only: Continuous infusion of a local anesthetic agent (bupivicaine 0.5%) intraarticularly only via Breg Pain Care 3000 Catheter
  Breg Pain Care 3000 Catheter: Pump that is designed to deliver local anesthetic directly to surgical site for several days.
Arm/Group | Intraartciularly Only | Patellar Tendon Harvest Site Only | Patellar Tendon Harvest Site and Intraarticular | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No